CLINICAL TRIAL: NCT04646993
Title: Which Decision After a First Venous Thromboembolism? The WHITE Study
Brief Title: WHITE Study: WHIch Decision After a First Venous ThromboEmbolism?
Acronym: WHITE
Status: Completed | Type: Observational
Sponsor: Arianna Anticoagulazione Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: WHITE_Final_20170920
Record Dates: First submitted 2020-11-18; First posted 2020-11-30 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2021-03

CONDITIONS: Venous Thromboembolism
Keywords: Deep vein thrombosis Anticoagulant Treatment; Lower limbs; Pulmonary embolism; Oral Anticoagulant Treatment
MeSH Terms: conditions — Venous Thromboembolism; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The WHITE study is a multicenter, multinational, investigators-initiated, observational, prospective study conducted in a consecutive series of ambulatory patients who had completed the recommended or practicable period of anticoagulation after a first-ever episode of venous thromboembolism (VTE)

The general aim of the study is to evaluate the distribution of decisions and of the reasons guiding the physician's decision on the modality to manage the secondary prevention of VTE in patients treated for a first-ever episode of VTE, after the initial 3-12 months of anticoagulant therapy.

DETAILED DESCRIPTION:
The WHITE study is an international, non-profit, multicenter, observational, prospective and no profit study 3,200 subjects having experienced a first-ever episode of DVT of the lower limbs and/or PE, receive anticoagulation therapy for a period as recommended by international and/or local practice guidelines will be enrolled across all the countries participating to the study.

When this recommended period expires, the attending physician has to decide whether to continue with anticoagulation, switch to anti-thrombotic of another class, or stop any prophylactic pharmacological treatment.

The primary objective of the study is the evaluation of the distribution of decisions and of the reasons guiding the physician's decision on the modality to manage the secondary prevention of VTE in patients treated for a first-ever episode of VTE, after the initial 3-12 months of anticoagulation therapy.

The secondary objective is the collection of data during the follow-up: the frequency of thromboembolic complications, of bleeding complications, or death from any cause.

ELIGIBILITY:
Inclusion Criteria:

1. subjects who provided a written informed consent and authorization for disclosure of protected health information;
2. male and female adult or elderly patients of any ethnicity having had a first-ever event of provoked or unprovoked DVT of the lower limbs and/or PE and treated with oral anticoagulant
3. for whom the center is in possession of all the data relevant to the index event;
4. having a permanent reference contact.

Exclusion Criteria:

1. subjects <18 years old;
2. subjects unable or unwilling to issue the written informed consent;
3. subjects for whom the information relevant to the index event are incomplete or inaccessible to the Investigator;
4. subject in whom the index event was a DVT not of the lower limbs;
5. subjects with life expectancy of less than 2 years;
6. subjects participating in any other clinical study, regardless of its nature;
7. subjects considered, by the attending physician, unable to comply with the study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients of any ethnicity having had a first-ever event of provoked or unprovoked DVT of the lower limbs and/or PE given maintenance anticoagulants (NOACs, VKAs, or LMWHs) according to the local procedures (usually for 3 to 12 months) and to be re-evaluated to decide the treatment to be prescribed after such period by the attending physicians
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Number of patients who continue or stop the anticoagulant treatment | From the end of the 3rd month to the end of 12th month of anticoagulant treatment
  Registration of number of patients who continue or stop the treatment; registration of type reasons guiding the attending physician's decision on the management of secondary prevention (eg: Bleeding score, laboratory test, presence of residual vein trombosis, risk or recurrence)

SECONDARY OUTCOMES:
Frequence of adverse events during follow-up | Frome the first day of enrollment up to 24 monhts
  the frequency of thromboembolic complications, of bleeding complications, or death from any cause monitored during the follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jiří Matuška, Prof, Study Director — Clinical Trial Centre, Hodonin, Czech Republic
Locations (1):
- Clinical Trial Centre, MATMED, Hodonín, Czechia

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/93/NCT04646993/Prot_SAP_000.pdf